CLINICAL TRIAL: NCT01075243
Title: A Study to Compare the Analgesic Efficacy of Two Different Paracetamol Doses as Measured by Post-operative Pain Relief
Brief Title: Post-operative Dental Pain Study Comparing Two Different Dosage of Analgesic Efficacy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4000685
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Post-surgical Dental Pain
Keywords: dental pain; paracetamol; Post-surgical dental pain
MeSH Terms: conditions — Toothache | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paracetamol 1000mg (Experimental): Paracetamol 1000mg
  Interventions: Drug: Paracetamol 1000 mg
- Paracetamol 650 mg (Experimental): Paracetamol 650 mg
  Interventions: Drug: Paracetamol 650 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol 1000 mg — Paracetamol 1000mg
  Arms: Paracetamol 1000mg
Drug: Paracetamol 650 mg — Paracetamol 650 mg
  Arms: Paracetamol 650 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
GlaxoSmithKline will be conducting this trial to compare analgesic efficacy of paracetamol 1000 mg vs 650 mg. The post-surgical dental pain model will be used to evaluate the analgesic efficacy of paracetamol. Each subject will be enrolled in the study for up to six weeks. The duration of the entire study will be approximately 18 weeks. Each subject will have to come to the clinic for three visits (Screening, Treatment and Follow up visits).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 45 years with moderate-to-severe dental pain as assessed by verbal rating scale (VRS) and confirmed by a score of at least 50 mm out of 100 mm using a visual analogue (VAS) following the surgical removal of up to two mandibular third molars. If only one mandibular third molar is removed, it must be a full bony impaction. If two mandibular third molars are removed, both may be partial bony impactions OR there may be a combination of one full bony impaction with the second tooth being erupted, soft tissue impaction, or partial bony impaction. Ipsilateral maxillary third molars may be removed at the surgeon's discretion, regardless of impaction level.

Exclusion Criteria:

* Pregnant and lactating females
* Allergy/intolerance to study materials or nitrous oxide or local anaesthetic used during surgery
* Current or recurrent liver, kidney or cardiac disease, stomach ulcers, gastrointestinal bleeding, gastroesophageal reflux disease, bronchospasm, rhinitis, urticaria or asthma

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 401 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Yue Y, Collaku A, Brown J, Buchanan WL, Reed K, Cooper SA, Otto J. Efficacy and speed of onset of pain relief of fast-dissolving paracetamol on postsurgical dental pain: two randomized, single-dose, double-blind, placebo-controlled clinical studies. Clin Ther. 2013 Sep;35(9):1306-20. doi: 10.1016/j.clinthera.2013.07.422. Epub 2013 Aug 22. PMID 23972577

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Of 722 screened participants, 321 were considered to be screen failures. Remaining 401 were randomized to study treatments.
Groups:
- Paracetamol Caplet 1000 Milligrams (mg): Participants were administered with two paracetamol fast dissolving (FD) 500 mg caplets (Total dose= 1000 mg), and two placebo standard paracetamol caplets with 150 milliliter (mL) of water through oral route.
- Paracetamol Caplet 650 mg: Participants were administered with two standard paracetamol 325 mg caplets (Total dose = 650 mg) and two placebo FD caplets, with 150 mL of water through oral route.
- Placebo Caplet: Participants were administered with two standard and two FD placebo caplets, with 150 mL of water through oral route.
Period: Overall Study
Arm/Group | Paracetamol Caplet 1000 Milligrams (mg) | Paracetamol Caplet 650 mg | Placebo Caplet
Started | 163 | 158 | 80
Completed | 157 | 155 | 80
Not Completed | 6 | 3 | 0
Not completed — Lost to Follow-up | 5 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Paracetamol Caplet 1000mg: Participants were administered with two paracetamol FD 500 mg caplets (Total dose= 1000 mg), and two placebo standard paracetamol caplets with 150 mL of water through oral route.
- Total: Total of all reporting groups
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet | Total
Number analyzed (Participants) | 163 | 158 | 80 | 401
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.7 (2.26) | 20.4 (2.81) | 20.6 (2.76) | 20.2 (2.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 104 | 56 | 262
  Male | 61 | 54 | 24 | 139
Number of participants with pain severity score measured on a rating scale [Number; unit: Participants] — Pain severity score was assessed on a 4-point categorical verbal rating scale. Total possible pain severity score range was no pain, mild pain, moderate and severe.
  Participants
    Moderate | 109 | 106 | 53 | 268
    Severe | 54 | 52 | 27 | 133

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Relief and Pain Intensity Differences From 0 to 6 Hours (SPRID 6 Hours)
Description: SPRID:Sum of Pain Intensity Difference (SPID) and Total Pain Relief (TOTPAR) at each post-dosing time-point. SPRID score ranged from -5.8 (least pain relief) to 40.3 (highest pain relief). SPID and TOTPAR were calculated as weighted sums of Pain Intensity Differences (PID) and Pain Relief Scores (PRS) at each measurement time, respectively. PID was derived by subtracting the pain severity score at a given post-dosing time-point from the baseline [pain severity score range:0-no pain, 1-mild pain, 2-moderate pain, 3-severe pain using a 4-point categorical Verbal Rating Scale (VRS)]. If the subject rated pain intensity as 2 or 3, pain was assessed using a 100 mm Visual Analog Scale (VAS) [0 (no pain), 100 (worst pain)]. VAS scores were converted into PID scores by subtracting them from baseline pain scores. PRS was assessed on 5-point categorical pain relief rating scale [0-no relief, 1-little relief, 2-some relief, 3-a lot of relief, 4-complete relief]
Time Frame: Every two hours from Baseline to 6 hours post dose
Population: Intent to Treat (ITT) population: All participants who received one study treatment and have at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
Score on a scale | 16.08 (10.68) | 12.42 (9.89) | 4.63 (8.82)
Statistical Analysis 1: Comparison: Paracetamol Caplet 1000mg vs Paracetamol Caplet 650 mg; Null hypothesis considered no difference in SPRID^6h between Paracetamol 1000 mg caplet and Paracetamol 650 mg caplet; Test type: Superiority or Other; p = 0.0009, ANCOVA; ANCOVA model included factors for treatment as a fixed effect and baseline assessment of pain intensity (VAS score) as a covariate; Adjusted Mean Difference = 3.71, 95% CI 2-sided [1.53 to 5.89] — Difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 2: Comparison: Paracetamol Caplet 1000mg vs Placebo Caplet; Null hypothesis considered no difference in SPRID^6h between Paracetamol 1000 mg caplet and placebo caplet; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Mean DIfference = 11.33, 95% CI 2-sided [8.66 to 14.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Paracetamol Caplet 650 mg vs Placebo Caplet; Null hypothesis considered no difference in SPRID^6h between Paracetamol 650 mg caplet and placebo caplet; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Mean Difference = 7.63, 95% CI [4.94 to 10.31] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Time to Confirmed First Perceptible Relief
Description: Participants recorded the time to first perceptible relief by starting the first stopwatch at the time of dosing and stopping it when he/she experienced the first perceptible pain relief. The first perceptible pain relief was confirmed if the participant also stopped the second stopwatch indicating meaningful relief.
Time Frame: Baseline to 6 hours post dose
Population: ITT population: All participants who received one study treatment and have at least one post-baseline efficacy assessment. Participants who did not achieve first perceptible pain relief during the 6 hours of the study period or took rescue medication were censored at the time 360 minutes.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
minutes | 54.72 (104.911) | 69.67 (120.501) | 225.70 (162.884)

3. Secondary Outcome: Time to Onset of Meaningful Pain Relief
Description: Participants recorded the time to meaningful relief by stopping a second stopwatch when they first began to experience meaningful relief.
Time Frame: Baseline to 6 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
minutes | 70.53 (101.474) | 88.16 (115.955) | 247.14 (143.028)

4. Secondary Outcome: Time to Start Using Rescue Medication
Description: Median time of use of rescue medication by participants.
Time Frame: Baseline to 6 hours post dose
Population: ITT population: All participants who received one study treatment and had at least one post-baseline efficacy assessment. Participants who did not achieve first perceptible pain relief during the 6 hours of the study period or took rescue medication were censored.
Measure: Median (Full Range); unit: minutes
Groups:
- Paracetamol Caplet 1000 mg: Participants were administered with two paracetamol FD 500 mg caplets (Total dose= 1000 mg), and two placebo standard paracetamol caplets with 150 mL of water through oral route.
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
minutes | 360.00 [124.00 to 360.00] | 314.00 [123.00 to 360.00] | 131.00 [115.00 to 360.00]

5. Secondary Outcome: Percentage of Participants Who Took Rescue Medication at 2 Hours
Description: Percentage of participants who received rescue medication at different time points post dose.
Time Frame: Baseline to 2 hours post dose
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
Percentage of participants | 0.00 | 0.00 | 1.30

6. Secondary Outcome: Percentage of Participants Who Took Rescue Medication at 6 Hours
Description: Percentage of participants who received rescue medication at different time points post dose.
Time Frame: Baseline to 6 hours post dose
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
Percentage of participants | 44.20 | 51.90 | 70.00

7. Secondary Outcome: SPRID at 2 Hours
Description: SPRID:Sum of Pain Intensity Difference (SPID) and Total Pain Relief (TOTPAR) at each post-dosing time-point. SPRID score ranged from -1.8 (least pain relief) to 12.3 (highest pain relief). SPID and TOTPAR were calculated as weighted sums of Pain Intensity Differences (PID) and Pain Relief Scores (PRS) at each measurement time, respectively. PID was derived by subtracting the pain severity score at a given post-dosing time-point from the baseline [pain severity score range:0-no pain, 1-mild pain, 2-moderate pain, 3-severe pain using a 4-point categorical Verbal Rating Scale (VRS)]. If the subject rated pain intensity as 2 or 3, pain was assessed using a 100 mm Visual Analog Scale (VAS) [0 (no pain), 100 (worst pain)]. VAS scores were converted into PID scores by subtracting them from baseline pain scores. PRS was assessed on 5-point categorical pain relief rating scale [0-no relief, 1-little relief, 2-some relief, 3-a lot of relief, 4-complete relief
Time Frame: Every two hours from baseline to 2 hours post dose
Population: All participants who received one study treatment and have at least one post-baseline efficacy assessment. Participants who did not achieve first perceptible pain relief during the 6 hours of the study period or took rescue medication were censored at the time 360 minutes.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
Score on a scale | 6.49 (3.11) | 5.57 (2.94) | 1.55 (2.45)

8. Secondary Outcome: SPRID at 4 Hours
Description: SPRID:Sum of Pain Intensity Difference (SPID) and Total Pain Relief (TOTPAR) at each post-dosing time-point. SPRID score ranged from -3.8 (least pain relief) to 26.3 (highest pain relief). SPID and TOTPAR were calculated as weighted sums of Pain Intensity Differences (PID) and Pain Relief Scores (PRS) at each measurement time, respectively. PID was derived by subtracting the pain severity score at a given post-dosing time-point from the baseline [pain severity score range:0-no pain, 1-mild pain, 2-moderate pain, 3-severe pain using a 4-point categorical Verbal Rating Scale (VRS)]. If the subject rated pain intensity as 2 or 3, pain was assessed using a 100 mm Visual Analog Scale (VAS) [0 (no pain), 100 (worst pain)]. VAS scores were converted into PID scores by subtracting them from baseline pain scores. PRS was assessed on 5-point categorical pain relief rating scale [0-no relief, 1-little relief, 2-some relief, 3-a lot of relief, 4-complete relief
Time Frame: Every two hours from baseline to 4 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
Score on a scale | 12.09 (6.93) | 9.45 (6.19) | 3.00 (5.27)

9. Secondary Outcome: Total Pain Relief Score (TOTPAR) at 2 Hours
Description: TOTPAR was calculated as sum of products of pain relief (PR) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0-15, 15-30, 30-45, 45-60, 60-90, 90-120. Higher score indicated greater pain relief.
  TOTPARt = ∑PR x (timet - timet-1).
  PR score was assessed at each of the above time-points based on a 5-point categorical scale [0-no relief, 1-little relief, 2-meaningful relief, 3-a lot of relief, 4-complete relief].
Time Frame: Every two hours from baseline to 2 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
Score on a scale | 4.31 (1.88) | 3.80 (1.89) | 1.36 (1.59)

10. Secondary Outcome: TOTPAR at 4 Hours
Description: TOTPAR was calculated as sum of products of pain relief (PR) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0-15, 15-30, 30-45, 45-60, 60-90, 90-120, 120-240. Higher score indicated greater pain relief.
  TOTPARt = ∑PR x (timet - timet-1).
  PR score was assessed at each of the above time-points based on a 5-point categorical scale [0-no relief, 1-little relief, 2-meaningful relief, 3-a lot of relief, 4-complete relief].
Time Frame: Every two hours from baseline to 4 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
Score on a scale | 8.21 (4.10) | 6.64 (3.97) | 2.79 (3.46)

11. Secondary Outcome: TOTPAR at 6 Hours
Description: TOTPAR was calculated as sum of products of pain relief (PR) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0-15, 15-30, 30-45, 45-60, 60-90, 90-120, 120-240, 240-300 and 300-360. Higher score indicated greater pain relief.
  TOTPARt = ∑PR x (timet - timet-1).
  PR score was assessed at each of the above time-points based on a 5-point categorical scale [0-no relief, 1-little relief, 2-meaningful relief, 3-a lot of relief, 4-complete relief].
Time Frame: Every two hours from baseline to 6 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
Score on a scale | 11.06 (6.41) | 8.83 (6.30) | 4.29 (5.80)

12. Secondary Outcome: Sum of Pain Intensity Difference (SPID) Scores at 2 Hours
Description: SPID was calculated as sum of products of Pain Intensity Differences (PID) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0-15, 15-30, 30-45, 45-60, 60-90, 90-120. Positive and higher scores indicate greater reduction in pain.
  SPIDt = ∑PID x (timet - timet-1)
  Pain Intensity was assessed at baseline and at each time-point based on a 4-point categorical Verbal Rating Scale (VRS) scale: 0-no pain, 1-mild pain, 2-moderate pain, 3-severe pain.
  If the subject rated pain intensity as "2" or "3", pain was assessed using a 100 mm Visual Analog Scale (VAS) [0 (no pain), 100 (worst pain)]. VAS scores were converted into PID scores by subtracting them from pain scores taken at baseline.
Time Frame: Every two hours from baseline to 2 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
Score on a scale | 2.17 (1.37) | 1.77 (1.20) | 0.19 (1.03)

13. Secondary Outcome: SPID Scores at 4 Hours
Description: SPID was calculated as sum of products of Pain Intensity Differences (PID) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0-15, 15-30, 30-45, 45-60, 60-90, 90-120, 120-240. Positive and higher scores indicate greater reduction in pain.
  SPIDt = ∑PID x (timet - timet-1)
  Pain Intensity was assessed at baseline and at each time-point based on a 4-point categorical Verbal Rating Scale (VRS) scale: 0-no pain, 1-mild pain, 2-moderate pain, 3-severe pain.
  If the subject rated pain intensity as "2" or "3", pain was assessed using a 100 mm Visual Analog Scale (VAS) [0 (no pain), 100 (worst pain)]. VAS scores were converted into PID scores by subtracting them from pain scores taken at baseline.
Time Frame: Every two hours from baseline to 4 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
Score on a scale | 3.88 (3.06) | 2.81 (2.52) | 0.20 (2.13)

14. Secondary Outcome: SPID Scores at 6 Hours
Description: SPID was calculated as sum of products of Pain Intensity Differences (PID) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0-15, 15-30, 30-45, 45-60, 60-90, 90-120, 120-240, 240-300 and 300-360. Positive and higher scores indicate greater reduction in pain.
  SPIDt = ∑PID x (timet - timet-1)
  Pain Intensity was assessed at baseline and at each time-point based on a 4-point categorical Verbal Rating Scale (VRS) scale: 0-no pain, 1-mild pain, 2-moderate pain, 3-severe pain.
  If the subject rated pain intensity as "2" or "3", pain was assessed using a 100 mm Visual Analog Scale (VAS) [0 (no pain), 100 (worst pain)]. VAS scores were converted into PID scores by subtracting them from pain scores taken at baseline.
Time Frame: Every two hours from baseline to 6 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
Score on a scale | 5.02 (4.63) | 3.59 (4.01) | 0.34 (3.51)

15. Secondary Outcome: Participants Global Assessment to Response to Treatment (PGART)
Description: PGART was measured by a score in a scale from 0-4: 0- Poor; 1- Fair 2- Good; 3- Very Good; 4- Excellent.
Time Frame: Baseline to 6 hours post dose
Population: ITT population: All participants who received study treatment and had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Number analyzed (Participants) | 163 | 158 | 80
Score on a scale | 2.20 (1.13) | 1.80 (1.18) | 0.80 (1.05)

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported following administration of any investigational product, or for up to 5 days after the last administration of investigational product were recorded.
Arm/Group | Paracetamol Caplet 1000mg | Paracetamol Caplet 650 mg | Placebo Caplet
Serious Adverse Events (participants affected / at risk) | 0/163 | 0/158 | 0/80
Other Adverse Events (participants affected / at risk) | 28/163 | 28/158 | 18/80
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paracetamol Caplet 1000mg (N=163) | Paracetamol Caplet 650 mg (N=158) | Placebo Caplet (N=80)
Nausea (Gastrointestinal disorders) | 17 (18) | 17 (17) | 7 (8)
Vomiting (Gastrointestinal disorders) | 7 (7) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 6 (6) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.